CLINICAL TRIAL: NCT07346222
Title: San Matteo Endocarditis Registry STEADY
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Elena Maria Seminari, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: STEADY
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Endocarditis Infective
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

SUMMARY:
The general objective of this study is to deepen the knowledge of patients affected by endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted from 1stJannary 2009 to 31 Dec 2029 to the Fondazione IRCCS Policlinico San Matteo with a diagnosis of IE according to modified Duke criteria

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a study conducted on the population affected by endocarditis admitted to the wards of our hospital and observational, i.e. having the sole aim of describing the characteristics of this type of critically ill patients.
Sampling Method: Non-Probability Sample
Enrollment: 418 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2030-11-13 (Estimated)

PRIMARY OUTCOMES:
describes the characteristics and clinical course that correlate with an adverse clinical outcome. | 2029

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy, Italy